CLINICAL TRIAL: NCT03935425
Title: FitMi Plus: Smart Functional Modules for Practicing Activities of Daily Living After Stroke
Brief Title: FitMi Plus Home Therapy for Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Flint Rehabilitation Devices, LLC (Industry)
Collaborators: University of California, Irvine (Other); Rancho Research Institute, Inc. (Other)
Responsible Party: Principal Investigator, Flint Rehabilitation Devices, LLC, Vice President, Flint Rehabilitation Devices, LLC
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1R44HD097803-01 (NIH)
Record Dates: First submitted 2019-04-25; First posted 2019-05-02 (Actual); Results first posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Cerebral Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- FitMi Plus (Experimental): Participants will perform targeted movement exercises by interacting with the FitMi Plus Functional modules at least 50% of the time they spend exercising.
  Participants will be asked to exercise at least 3 hours per week for 3 consecutive weeks.
  Interventions: Device: FitMi Plus
- FitMi Basic (Active Comparator): Participants will perform targeted movement exercises by interacting with the FitMi Basic pucks, as described and monitored on a computer.
  Participants will be asked to exercise at least 3 hours per week for 3 consecutive weeks.
  Interventions: Device: FitMi Basic

INTERVENTIONS:
Device: FitMi Plus — A set of common objects that couple with a wireless sensor platform to allow the performance of functional exercises to be measured by a motivating software platform.
  Arms: FitMi Plus
Device: FitMi Basic — A wireless sensor platform that allows movement subcomponents and point-to-point exercises to be measured by a motivating software platform.
  Arms: FitMi Basic

SUMMARY:
The investigators will investigate the efficacy of a newly developed functional exercise device (FitMi Plus) for people in the chronic stage after a stroke compared to the FitMi Basic (i.e. without functional exercises). FitMi Plus combines objects commonly used during activities of daily living with sensors that can track and record the patient's direction and degree of movement as they perform specific functional tasks described on a computer.

ELIGIBILITY:
Inclusion Criteria:

* Experienced 1 or more strokes >6 months prior to enrollment
* Upper Extremity Fugl-Meyer Score >=15 and <=55 out of 66
* Absence of moderate to severe upper extremity pain (<= 4 out of 10 on the visual-analog pain scale)
* Ability to understand the instructions to operate FitMi products

Exclusion Criteria:

* Lack of concurrent severe medical problems
* Lack of visual deficits
* Lack of severe neglect or apraxia
* No concurrent enrollment in another therapy study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-11-29 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Reinkensmeyer, PhD, Principal Investigator — University of California, Irvine; Susan Shaw, MD, Principal Investigator — Rancho Research Institute, Inc.
Locations (2):
- United States (2):
  - Rancho Research Institute, Inc, Downey, California
  - Human Neuroperformance Laboratory at University of California Irvine, Irvine, California

RESULTS

PARTICIPANT FLOW:
Groups:
- FitMi Plus: Participants will perform targeted movement exercises by interacting with the FitMi Plus Functional modules at least 50% of the time they spend exercising.
  Participants will be asked to exercise at least 3 hours per week for 3 consecutive weeks.
  FitMi Plus: A set of common objects that couple with a wireless sensor platform to allow the performance of functional exercises to be measured by a motivating software platform.
- FitMi Basic: Participants will perform targeted movement exercises by interacting with the FitMi Basic pucks, as described and monitored on a computer.
  Participants will be asked to exercise at least 3 hours per week for 3 consecutive weeks.
  FitMi Basic: A wireless sensor platform that allows movement subcomponents and point-to-point exercises to be measured by a motivating software platform.
Period: Overall Study
Arm/Group | FitMi Plus | FitMi Basic
Started | 25 | 25
Completed | 24 | 24
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FitMi Plus | FitMi Basic | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.4 (14.7) | 54.0 (13.0) | 55.2 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 14
  Male | 17 | 19 | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 12 | 25
  Not Hispanic or Latino | 8 | 13 | 21
  Unknown or Not Reported | 4 | 0 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 6 | 3 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 1 | 5
  White | 7 | 9 | 16
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 8 | 12 | 20

OUTCOME MEASURES:

1. Primary Outcome: Change in Motor Activity Log
Description: A self-reported measure of the quality of movement and amount of use of the impaired upper extremity across a set of activities of daily living. Minimum value = 0, maximum value = 5, higher scores = better outcome
Time Frame: Baseline and One-Month Post-Treatment, at seven weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FitMi Plus | FitMi Basic
Number analyzed (Participants) | 24 | 24
score on a scale
  Amount of Use | 0.60 (0.53) | 0.40 (0.39)
  Quality of Movement | 0.64 (0.48) | 0.44 (0.35)
Statistical Analysis 1: Comparison: FitMi Plus vs FitMi Basic; Test type: Superiority; p = 0.11, t-test, 2 sided

2. Secondary Outcome: Change in Upper Extremity Fugl-Meyer
Description: A standardized assessment of arm impairment based on scores of 0-2 on 33 different tasks. Minimum value = 0, maximum value = 66, higher scores = better outcome
Time Frame: Baseline and One-Month Post-Treatment, at seven weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FitMi Plus | FitMi Basic
Number analyzed (Participants) | 25 | 25
score on a scale | 2.0 (3.3) | 1.0 (2.8)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from enrollment to one-month post-therapy, approximately 7 weeks.
Arm/Group | FitMi Plus | FitMi Basic
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-12-31): https://cdn.clinicaltrials.gov/large-docs/25/NCT03935425/Prot_SAP_002.pdf
  • Informed Consent Form (2021-04-20): https://cdn.clinicaltrials.gov/large-docs/25/NCT03935425/ICF_001.pdf